CLINICAL TRIAL: NCT03469973
Title: Partial Adenoidectomy in Cases of Velopharyngeal Dysfunction
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Basem Makram, Principal investigator, Assiut University
Other Study IDs: BASEMM
Record Dates: First submitted 2018-03-12; First posted 2018-03-19 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Velopharyngeal Insufficiency; Velopharyngeal Incompetence Due to Cleft Palate
MeSH Terms: conditions — Velopharyngeal Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Partial adenoidectomy — The procedure will be completely visualized with a 45 degrees, 4- mm nasal endoscope; the upper part of the adenoid will be removed using the microdebrider, while the lower part will be preserves to maintain the velopharyngeal competence.
  • Adenoid enlargement causing Obstructive Sleep-Disordered Breathing (OSDB) with velopharyngeal insufficiency (proved or suspected).

SUMMARY:
The velopharyngeal valve is a tridimensional muscular valve that is located between the oral and nasal cavities. It consists of the lateral and posterior pharyngeal walls as well as the soft palate. The role of the velopharyngeal valve is to separate the oral and nasal cavities during speech and swallowing.

DETAILED DESCRIPTION:
Velopharyngeal dysfunction is the inability to separate the oral and nasal cavities adequately during speech production through the actions of the velum and pharynx. Velopharyngeal dysfunction can be caused due to lack of tissue (velopharyngeal insufficiency) or lack of proper movement (velopharyngeal incompetence) of the walls. While Velopharyngeal dysfunction is commonly associated with cleft lip and palate, it can also be seen with submucous cleft and other noncleft conditions such as ablative palatal lesions, adenoidectomy, deafness or hearing loss, and cerebral palsy. In Velopharyngeal dysfunction, the incompletely closed velopharyngeal valve causes an inability to effectively manage the air stream for continuous speech causing hypernasal speech.

Adenoid hypertrophy may play a role in velopharyngeal closure especially in patients with palatal abnormality.

In 1958, Gibb indicated an incidence of hypernasality postadenoidectomy in approximately 1 of 2000 cases. Closure pattern of velopharyngeal valve in typical patients is velo-adenoidal rather than velopharyngeal closure. Adenoid mass is vital to velopharyngeal closure in such patients and removal necessitates a change in the pattern of velopharyngeal valving.

Trans-oral endoscopic partial (superior) adenoidectomy adenoidectomy enables the surgeon to inspect the velopharyngeal valve during the procedure; thus avoiding occurrence of velopharyngeal dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Adenoid enlargement causing Obstructive Sleep-Disordered Breathing (OSDB) with velopharyngeal insufficiency (proved or suspected).

Exclusion Criteria:

* Patients who had undergone any secondary corrective surgery for velopharyngeal insufficiency.
* Patients with craniofacial anomalies.
* Any associated medical comorbidity that contraindicates general anesthesia.
* Refusal of enrollment in the research by the patients or care givers.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will be conducted on Otorhinolaryngology Department, Assiut University Hospital, in the period between 1⁄5∕2018 and 1∕5⁄2020.
  The study will be carried on 40 consecutive cases.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
40 patients diagnosed by velopharyngeal insufficiency will go for partial adenoidectomy completely visualised by 45 degrees, 4 mm nasal endoscope. The adenoid will be removed by using microdeprider. | Up to 2 years